CLINICAL TRIAL: NCT06481475
Title: A Randomized Double-blind Vehicle-controlled Parallel-dose Phase II Study Evaluating the Safety and Efficacy of a Recombinant Botulinum Neurotoxin Type a Injection (YY003) for the Treatment of Moderate to Severe Glabellar Lines in Adults
Brief Title: A Study to Investigate the Safety and Efficacy of YY003 in Adults with Moderate to Severe Glabellar Lines
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chongqing Claruvis Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YY003-001-US01
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Moderate to Severe Glabellar Lines
Keywords: YY003; Botulinum Toxin; Glabellar Lines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low dose YY003 (Experimental): Participants will receive a single dose over 5 injection sites on Day 1.
  Interventions: Biological: YY003
- High dose YY003 (Experimental): Participants will receive a single dose over 5 injection sites on Day 1.
  Interventions: Biological: YY003
- Vehicle control (Placebo Comparator): Participants will receive a single dose over 5 injection sites on Day 1.
  Interventions: Biological: Vehicle Control

INTERVENTIONS:
Biological: YY003 — Single treatment, intramuscularly injected into five sites. The total injection volume is 0.25 ml, 0.05 ml per site.
  Arms: High dose YY003; Low dose YY003
Biological: Vehicle Control — Single treatment, intramuscularly injected into five sites. The total injection volume is 0.25 ml, 0.05 ml per site.
  Arms: Vehicle control

SUMMARY:
The study is a two-part (Part A and Part B) randomized double-blind vehicle-controlled multi-center study in a total of 174 participants with moderate to severe glabellar lines. The objective of this study is to test the safety, efficacy, immunogenicity of YY003, and compare to vehicel control, in improving the appearance of moderate to severe glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

1. Participants (male or female) must be ≥18 years old, at the time of signing the informed consent.
2. At screening and baseline, participants must have moderate to severe glabellar lines at maximum frown (grade 2 or 3 on the relevant 4-point scale), as assessed by both the investigator and the participant.
3. Male or female (inclusive of all gender identities) participants are eligible to participate if they agree to practice adequate contraceptive methods during the study period and for at least 3 months after the study drug administration. Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
4. Participant must provide signed informed consent, including compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
5. Participant must have the time and ability to complete the study and comply with instructions, at the discretion of the investigator.

Exclusion Criteria:

1. Known allergy or hypersensitivity to any components of the investigational product or any botulinum toxin serotype.
2. A history or presence of ptosis, significant facial asymmetry, excessive dermatochalasis at screening or baseline.
3. A history or presence of facial nerve palsy at screening or baseline.
4. A positive HIV, hepatitis B or hepatitis C test at screening.
5. History or presence of other concomitant diseases which are assessed by the investigator to be unsuitable for participation in this clinical research.
6. History of drug or alcohol abuse.
7. History or presence of epilepsy.
8. Have a serious mental disorder that, in the Investigator's opinion, may affect participant compliance with the study.
9. Female who is pregnant or breast feeding.
10. Abnormal laboratory tests that, in the Investigator's assessment, are not appropriate for participation in this study.
11. Participation in an investigational device or drug study within 30 days or 5 half-lives (whichever is longer) prior to screening.
12. Study center personnel, close relatives of the study center personnel, employees or close relatives of employees at the sponsor company.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Satety: Incidence of treatment-emergent adverse events (TEAEs), adverse events of special interest (AESI), and serious adverse events (SAEs) | within 4 weeks post-treatment
Efficacy: The proportion of participants achieving a score of 0 or 1 and at least a two-grade improvement from baseline, on both the investigator's assessment and the participant's self-assessmenti of glabellar line severity at maximum frown | at Week 4 post-treatment visit

SECONDARY OUTCOMES:
Incidence of anti-drug antibodies and neutralizing antibodies | Within 12 Weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - St George Dermatology & Skin Cancer Centre, Sydney, New South Wales
  - Skin Health Institute, Melbourne, Victoria
  - Dermatology Institute of Victoria, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No